CLINICAL TRIAL: NCT02207582
Title: Prefrontal Transcranial Random Noise Stimulation in Patients With Depression
Acronym: tRNS-depr
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no efficacy
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., MD, PhD, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tRNS in depression
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Depression
Keywords: depression; trns
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum Prefrontal tRNS (Experimental): 2mA of tRNS (DC-Stimulator, NeuroConn GmbH, Germany) with a zero offset will be applied to the left and right dorsolateral prefrontal cortex. Treatment will consist of 15 days with 20 minutes stimulation per day. Voltage will be ramped at the begin and end of a stimulation for 10 seconds.
  Interventions: Device: Verum Prefrontal tRNS
- Placebo Prefrontal tRNS (Placebo Comparator): 2mA of tRNS (DC-Stimulator, NeuroConn GmbH, Germany) with a zero offset will be applied to the left and right dorsolateral prefrontal cortex. Treatment will consist of 15 days with 20 minutes stimulation per day. Voltage will be ramped at the begin and end of a stimulation for 10 seconds. Placebo stimulation will consist of just applying the ramps at the begin and end of the stimulation.
  Interventions: Device: Placebo Prefrontal tRNS

INTERVENTIONS:
Device: Verum Prefrontal tRNS — 2mA of tRNS (DC-Stimulator, NeuroConn GmbH, Germany) with a zero offset will be applied to the left and right dorsolateral prefrontal cortex. Treatment will consist of 15 days with 20 minutes stimulation per day. Voltage will be ramped at the begin and end of a stimulation for 10 seconds.
  Arms: Verum Prefrontal tRNS
Device: Placebo Prefrontal tRNS — 2mA of tRNS (DC-Stimulator, NeuroConn GmbH, Germany) with a zero offset will be applied to the left and right dorsolateral prefrontal cortex. Treatment will consist of 15 days with 20 minutes stimulation per day. Voltage will be ramped at the begin and end of a stimulation for 10 seconds. Placebo stimulation will consist of just applying the ramps at the begin and end of the stimulation.
  Arms: Placebo Prefrontal tRNS

SUMMARY:
Transcranial random noise stimulation is used to stimulate the prefrontal cortices in patients with depression. It's a placebo-controlled two-arm study.

DETAILED DESCRIPTION:
Transcranial random noise stimulation (tRNS) is a non-invasive electric stimulation technique of the brain which was shown to be superior effective in contrast to other electric stimulation such as transcranial direct current stimulation (tDCS). These studies investigated mainly healthy controls and specific tasks. Only one case report is available for depression. Here we stimulate patients with depression with tRNS in a placebo-controlled two-arm design. Stimulation will be done as add-on to standard therapy. Electrodes will be applied over both dorsolateral prefrontal cortices which are standard target points of tDCS and also transcranial magnetic stimulation in depression.

ELIGIBILITY:
Inclusion Criteria:

* episode of depression (unipolar or bipolar) ( ICD-10)
* female or male between 18 and 70 years old
* skills to participate in all study procedures
* 18 or more points in the Hamilton rating scale or depression
* written informed consent

Exclusion Criteria:

* clinically relevant unstable internal or neurological comorbidity
* evidence of significant brain malformations or neoplasm, head injury
* cerebral vascular events
* neurodegenerative disorders affecting the brain or prior brain surgery
* metal objects in and around body that can not be removed
* pregnancy
* alcohol or drug abuse
* eczema on the head
* heart pacemaker
* high dose tranquillizers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10-14 (Actual); Study Completion 2016-12-06 (Actual)

PRIMARY OUTCOMES:
Change in depression severity measured by the 21-item Hamilton Depression Rating Scale (baseline (-day 3) versus end of treatment (day 19)) | day 3; day 19
  Change in depression severity measured by the 21-item Hamilton Depression Rating Scale (baseline (-day 3) versus end of treatment (day 19))

SECONDARY OUTCOMES:
Change in depression severity measured by the Major Depression Inventory over the course of the trial | day 10; -day 3; day 5; day 12; day 19; day 75
  Change in depression severity measured by the Major Depression Inventory over the course of the trial
Number of responders (response = decrease of the Hamilton Depression rating scale for at least 50%) (baseline versus end of treatment) | day 3; day 19
  Number of responders (response = decrease of the Hamilton Depression rating scale for at least 50%) (baseline versus end of treatment)
Change in the Clinical Global Impression Scale over the course of the trial | day 3; day 5; day 12; day 19; day 75
  Change in the Clinical Global Impression Scale over the course of the trial
Change in the Beck Depression Inventory over the course of the trial | day 3; day 5; day 12; day 19; day 75
  Change in the Beck Depression Inventory over the course of the trial
Change in alertness, working memory and divided attention over the course of the trial | day 3; day 19; day 75
  Change in alertness, working memory and divided attention over the course of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, Principal Investigator — University of Regensburg
Locations (1):
- University of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No